CLINICAL TRIAL: NCT06695741
Title: Reduced Dose of Cyclophosphamide Combined With Standard Immunosuppressive Therapy as Front-line Therapy in Patients With Severe Aplastic Anemia
Brief Title: Reduced Dose of Cyclophosphamide Combined With Standard Immunosuppressive Therapy to Treat Severe Aplastic Anemia
Acronym: hypo-CASH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Jun Shi, Director of the Red Blood Cell Disorders Center & Director of the Regenerative Medicine Clinic, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hypo-CASH-2024
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Severe Aplastic Anemia; Cyclophosphamide Reduced-dose; Immunosuppressive Therapy
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypo-CASH (Experimental): ALG/CsA and herombopag and reduced dose of cyclophosphamide
  Interventions: Drug: Reduced dose of cyclophosphamide combined with standard immunosuppressive therapy

INTERVENTIONS:
Drug: Reduced dose of cyclophosphamide combined with standard immunosuppressive therapy — Severe aplastic anemia patients will receive a daily dose of Anti-lymphocyte globulin (25mg/kg) for the initial five days at the beginning of the treatment. Cyclosporine will be administered daily at a dosage of 3-5mg/kg. Herombopag will be administered daily at a dosage of 15mg starting from the first day of treatment and continuing for a duration of six months. Cyclophosphamide (20mg/kg) will be administered on days 15-16.

SUMMARY:
This is a prospective, single-center, single-arm, phase 2 study. This study aims to evaluate the efficacy and safety of anti-lymphocyte globulin plus herombopag in combination with the reduced dose of cyclophosphamide (hypo-CASH) for severe aplastic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of naïve severe or very severe aplastic anemia
* Male or female age ≥ 12 years
* Unwilling or unable to receive allogeneic hematopoietic stem cell transplantation.
* ECOG performance status ≤2
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* Previously received immunosuppressive therapy > 4 weeks
* Previously treated with TPO-RA > 4 weeks
* Have an allergy or intolerance to anti-lymphocyte globulin, cyclosporine, herombopag or cyclophosphamide.
* Uncontrolled fungal, bacterial, or viral infection. Hepatitis-associated aplastic anemia is allowed; hepatitis B or C infection is permitted unless it causes severe liver failure.
* Tested positive for HIV or syphilis
* Presence of severe liver, kidney, or heart failure, or other life-threatening comorbidities.
* History of radiotherapy and chemotherapy for malignant solid tumors in recent 5 years
* Combined with other serious disorders
* Pregnant or breast-feeding patients
* Patients considered to be ineligible for the study by the investigator for reasons other than the above.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Within 3 months
  Percentage of patients with hematological response. Hematological response includes complete rate, near complete rate(CR), very good partial response(VGPR), good partial response(GPR) and partial response(PR).

SECONDARY OUTCOMES:
Superior response rate | With in 6 months
  Percentage of patients with superior response, including CR, VGPR and GPR.
Overall response rate | With in 6 months
  Percentage of patients with hematological response. Hematological response includes complete rate, near complete rate(CR), very good partial response(VGPR), good partial response(GPR) and partial response(PR).
Incidence of the adverse event | Within 6 months
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event
Time to achieve robust superior response | Within 6 months
First time to response | Within 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Red Blood Cell Disorders Center and Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No